CLINICAL TRIAL: NCT03492970
Title: Characterization of Behavioral Disorders and 24 H-melatonin Level in Adults With Smith Magenis Syndrome
Brief Title: Melatonin in Adults With SMS
Acronym: SMS-adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hôpital le Vinatier (Other)
Collaborators: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2017-A02299-44
Record Dates: First submitted 2018-03-01; First posted 2018-04-10 (Actual); Last update posted 2019-04-22 (Actual); Status verified 2019-04

CONDITIONS: Smith Magenis Syndrome
MeSH Terms: conditions — Smith-Magenis Syndrome

STUDY DESIGN:
Intervention Model Description: To specify the evolution of the nycthéméral cycle of the secretion of melatonin in 10 adult subjects carrying a SMS
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 10 adult patients with SMS (Other): Specify the evolution of the nycthemeral cycle of melatonin secretion in adult subjects carrying an SMS Behavioral characterization of adult subjects with SMS Make recommendations on the management of sleep / sleep rhythm disorders and behavior in adult subjects with SMS
  Interventions: Biological: Hourly dosing of the nychtemeral secretion of melatonin

INTERVENTIONS:
Biological: Hourly dosing of the nychtemeral secretion of melatonin — Hourly dosing of the nychtemeral secretion of melatonin links and with sleep disorders and behavior of adult patients with SMS

SUMMARY:
Sleep-Wake and behavioral disorders in Smith Magenis Syndrome (SMS) are strongly linked to an inversion of the nychtemeral secretion of melatonin. This inversion have been described in children with SMS. However its evolution during adulthood remains unknown. The aim of this study is to assess 24hours melatonin levels in 10 adults with SMS in order to optimize medication in adults with SMS

DETAILED DESCRIPTION:
SMS is one of the rare syndromes in which the inversion of melatonin secretion is regular, which is an exceptional situation for the study of the influence of genetic factors on the regulation of sleep / wake rhythm. Recently, point mutations of the RAI1 gene (Retinoic Acid Induced 1) have been identified in individuals with the clinical features of SMS with a reversal of the secretion rate of melatonin ,highlighting the role of RAI1 in SMS sleep disorders.

Daytime secretion of melatonin is associated with significant drowsiness and plays a major role in diurnal behavior disorders, especially in younger people. Conversely, the absence of nocturnal melatonin is a causal factor in the shortening and fragmentation of nocturnal sleep .

Basically, little is known about the mechanisms that explain the inversion of the secretion rate of melatonin in SMS.

These aspects, and in particular the nycthemeral reversal of the melatonin cycle, have been described in a population of children and we do not know how these disturbances evolve in adulthood

ELIGIBILITY:
Inclusion Criteria:

* Patient with Smith Magenis Syndrome aged 18 years or older
* subject or guardian having signed the consent

Exclusion Criteria:

* Pregnant women
* Minor subject
* Diagnosis of Smith Magenis syndrome not certain
* Taking benzodiazepines or related substances
* Taking betablockers
* Major behavioral disorders versus indicating participation in this study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-03-07 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-03-30 (Actual)

PRIMARY OUTCOMES:
24h melatonin levels | 24 hours
  Plasmatic melatonin level will be assessed every hour during 24h for each subject

SECONDARY OUTCOMES:
Analysis of actimetry | 15 days
  At the end of the Visit 1 interview, an actimeter will be given to the patient to be worn on the previous two weeks before Visit 2. This will allow the evaluation of the sleep / wake rhythm in the usual life situation. The actimeter will be reported by the patient during the second visit .

CONTACTS AND LOCATIONS:
Overall Officials: POISSON ALICE, PH, Principal Investigator — CH LE VINATIER
Locations (1):
- CH Le Vinatier, Bron, Auvergne-Rhône-Alpes, France

IPD SHARING:
Plan to Share IPD: No